CLINICAL TRIAL: NCT00686439
Title: HUM 06-087: Proof of Concept Study : Adalimumab for the Treatment of Osteoarthritis
Brief Title: Adalimumab for Inflammatory Osteoarthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Walter Maksymowych, F.R.C.P.(C),Professor of Medicine, Consultant Rheumatologist, University of Alberta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM 06-087
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; adalimumab; mri
MeSH Terms: conditions — Osteoarthritis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adalimumab (Experimental)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — subcutaneous injection 40mg on alternate weeks
  Other Names: Humira
Drug: adalimumab — subcutaneous injection 40mg every other week
  Other Names: Humira

SUMMARY:
We will conduct a pilot study of the effectiveness of adalimumab for inflammatory osteoarthritis.

DETAILED DESCRIPTION:
This is a 20 patient pilot open-label study of the efficacy of adalimumab in inflammatory osteoarthritis of the knee. Primary endpoint is at 12 weeks and primary outcome is the OARSI responder index.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 40 years of age or older.
* If female, patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control: condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD) contraceptives (oral or parenteral) for three months prior to study drug administration),a vasectomized partner, total abstinence from sexual intercourse
* If patient is female and of childbearing potential, the results of a serum pregnancy test performed at Screening, prior to the first dose of adalimumab, must be negative.
* Patient has a diagnosis of OA of the index knee according to American College of Rheumatology criteria, including radiological evidence of OA (Kellgren-Lawrence grades 2 or 3).
* Patient has had continual pain for at least 6 months prior to inclusion in the study. This includes pain that has persisted despite conventional treatment, defined as any one of the following medications taken daily during the preceding month:acetaminophen (2- 4 grams per day)maximum tolerated and recommended doses of an NSAID, acetaminophen/codeine combination (i.e. Tylenol No 2, 3, 4) taken at least 3 times daily
* Patient has had daily knee pain for the month preceding study enrolment.
* Patient has a summed pain score of 125-400mm (visual analog scale) on the WOMAC pain sub-scale in the index (more symptomatic) knee.
* Patient has clinical evidence of a knee effusion in the index (more symptomatic) knee at Screening and Baseline.

Exclusion Criteria:

* Subject has a history of an allergic reaction or significant sensitivity to constituents of Adalimumab.
* Patient has a history of proven systemic arthritis such as rheumatoid arthritis.
* Patient has a concurrent medical or arthritic condition that could confound evaluation of the index joint e.g. post-traumatic or any secondary form of knee OA
* Patient has predominant patellofemoral disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
OARSI/OMERACT response | 12 weeks

SECONDARY OUTCOMES:
WOMAC Patient Global MRI | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: walter p maksymowych, FRCP, Principal Investigator — University of Alberta
Locations (1):
- The University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Maksymowych WP, Russell AS, Chiu P, Yan A, Jones N, Clare T, Lambert RG. Targeting tumour necrosis factor alleviates signs and symptoms of inflammatory osteoarthritis of the knee. Arthritis Res Ther. 2012 Oct 4;14(5):R206. doi: 10.1186/ar4044. PMID 23036475